CLINICAL TRIAL: NCT05024045
Title: A Phase 1 Study of Oral LOXO-338, a Selective BCL-2 Inhibitor, in Patients With Advanced Hematologic Malignancies
Brief Title: Study of Oral LOXO-338 in Patients With Advanced Blood Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18258; 2021-000060-30 (EudraCT Number); J3N-OX-JZRA (Other: Eli Lilly and Company); LOXO-BCL-20001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-cell Marginal Zone; Lymphoma, Non-Hodgkin; Multiple Myeloma; B-cell Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell
Keywords: BTKi; Hematologic disease; Small lymphocytic lymphoma; BCL-2 inhibitor; CLL; SLL; NHL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Mantle-Cell; Hematologic Diseases | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LOXO-338 (Monotherapy) (Experimental): LOXO-338 administered orally.
  Interventions: Drug: LOXO-338
- LOXO-338 + Pirtobrutinib (Combination) (Experimental): LOXO-338 administered orally in combination with pirtobrutinib
  Interventions: Drug: LOXO-338; Drug: Pirtobrutinib

INTERVENTIONS:
Drug: LOXO-338 — Oral
  Other Names: LY3847429
Drug: Pirtobrutinib — Oral
  Other Names: LOXO-305; LY3527727
  Arms: LOXO-338 + Pirtobrutinib (Combination)

SUMMARY:
The purpose of this study is to find out whether the study drug, LOXO-338, is safe and effective in patients with advanced blood cancer. Patients must have already received standard therapy. The study may last up to approximately 3 years.

DETAILED DESCRIPTION:
This study will be conducted in 2 parts. Part 1 will evaluate LOXO-338 as monotherapy. If safety and initial evidence of efficacy of LOXO-338 monotherapy are confirmed, part 2 will evaluate the combination of LOXO-338 with the highly selective, noncovalent Bruton's tyrosine kinase (BTK) inhibitor, pirtobrutinib (LOXO-305).

ELIGIBILITY:
Inclusion Criteria:

* B-cell malignancy.
* Patients must have received prior therapy.
* Patients must have an objective indication for therapy.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1.
* Anticipated life expectancy of greater than or equal to (≥) 12 weeks.
* Adequate bone marrow function.
* Adequate hepatic function.
* Creatinine clearance of ≥ 60 milliliters (mL)/minute.
* Ability to swallow tablets.
* Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation.
* Prior treatment-related adverse events (AEs) must have recovered to grade less than or equal to (≤) 1 or pretreatment baseline, with the exception of alopecia.
* Men with partners of childbearing potential or women of childbearing potential (WOCBP) must agree to use highly effective birth control.
* WOCBP must not be pregnant.
* Additional Inclusion Criteria for Patients with AL Amyloidosis

  * In Part 1 Dose Expansion, patients with AL amyloidosis are eligible based on prior detection of primary systemic light-chain amyloidosis.
  * Must have measurable disease of AL amyloidosis.
  * Prior local fluorescence in-situ hybridization (FISH) testing results for t(11;14) are required to be submitted prior to enrollment.

Exclusion Criteria:

* Prior to identification of an appropriate RP2D (Dose Expansion) of LOXO-338, a history of known, active or suspected:

  * Richter's transformation to diffuse large B-cell lymphoma (DLBCL), prolymphocyticleukemia, or Hodgkin lymphoma
  * Transformed low grade lymphoma
  * Burkitt or Burkitt-like lymphoma
  * Diffuse large B-cell lymphoma
  * AL amyloidosis
  * Multiple myeloma
  * Lymphoblastic lymphoma or leukemia
  * Posttransplant lymphoproliferative disorder
* Known or suspected history of central nervous system (CNS) involvement.
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor-modified T cell (CAR-T) therapy within the past 60 days and with any of the following:

  * Active graft versus host disease (GVHD)
  * Cytopenias from incomplete blood cell count recovery post-transplant or CAR-T therapy
  * Need for anti-cytokine therapy for toxicity from CAR-T therapy; residual symptoms of neurotoxicity Grade > 1 from CAR-T therapy
  * Ongoing immunosuppressive therapy
* Known human immunodeficiency virus (HIV) positive, regardless of cluster of differentiation 4 (CD4) count. Unknown or negative status eligible.
* Inability to take necessary uric acid lowering agents (i.e., allopurinol, rasburicase, orfebuxostat).
* Concurrent anticancer therapy.
* Concurrent treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers that can include antifungals.
* Use of ≥ 20 milligrams (mg) prednisone once a day (QD) or equivalent dose of steroid per day, within 7 days of start of study treatment. Patients may not be on any dose of prednisone intended for antineoplastic use.
* Vaccination with a live vaccine within 28 days prior to start of study therapy.
* Major surgery within four weeks of planned start of study therapy Prolongation of the QT interval corrected by Fridericia's Formula for heart rate (QTcF) greater than (>) 470 milliseconds (msec).
* Clinically significant cardiovascular disease.
* Female patient who is pregnant or lactating.
* Active second malignancy which may preclude assessment of DLT.
* Clinically significant active malabsorption syndrome including surgical resection of small intestine or other condition likely to affect gastrointestinal (GI) absorption of the orally administered study drugs.
* Active hepatitis B or C infection.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal) or other clinically significant active disease process.
* Active uncontrolled auto-immune cytopenia.
* Additional Exclusion Criteria for Patients with AL Amyloidosis (Part 1 Dose-Expansion)

  * Previous or current diagnosis of symptomatic MM.
  * Heart failure that, in the opinion of the Investigator, is on the basis of ischemic heart disease.
  * Supine systolic blood pressure < 90 mmHg, or symptomatic orthostatic hypotension in the absence of volume depletion.
  * N-terminal pro hormone natriuretic peptide (NT-proBNP) > 8500 ng/L (or BNP > 700 ng/L if NT-proBNP is not available by local or central testing).
* Additional exclusion criteria for patients enrolled to part 2: LOXO-338 and pirtobrutinib combination

  * Prior progression or intolerance to pirtobrutinib.
  * Patients requiring therapeutic anticoagulation with warfarin.
  * Known hypersensitivity to any component or excipient of pirtobrutinib.
  * In patients with history of myocardial infarction or congestive heart failure, documented left ventricular ejection fraction (LVEF) by any method of ≤ 45 percent (%) in the 12 months prior to planned start of study treatment.
  * History of uncontrolled or symptomatic arrhythmias including grade ≥ 3 arrhythmia on a prior BTK inhibitor.
  * History of major bleeding on a prior BTK inhibitor.
  * Current treatment with strong permeability glycoprotein (P-gp) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Part 1 - To determine the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of oral LOXO-338 | Cycle 1 (28 Days)
  Measured by the number of patients with dose-limiting toxicities (DLTs)
Part 1 - To determine the effect of LOXO-338 on response rates | Estimated up to 2 years
  Measured by the appropriate disease specified response criteria as appropriate to tumor type
Part 2 - To determine the safety and tolerability of LOXO-338 when given in combination with pirtobrutinib | Cycle 2 (28 Days)
  Measured by the number of patients with dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Part 1 - To characterize the pharmacokinetics (PK) properties of LOXO-338: Area under the plasma concentration versus time curve (AUC) | Predose up to 24 hours postdose
  PK: AUC of LOXO-338
Part 1 - To characterize the PK properties of LOXO-338: Maximum drug concentration (Cmax) | Predose up to 24 hours postdose
  PK: Cmax of LOXO-338
Part 1 - To assess preliminary antitumor activity of LOXO-338 based on overall response rate (ORR) | Estimated up to 2 years
  ORR
Part 1 - To assess preliminary antitumor activity of LOXO-338 based on progression-free survival (PFS) | Estimated up to 2 years
  PFS
Part 1 - To assess preliminary antitumor activity of LOXO-338 based on time-to-progression (TTP) | Estimated up to 2 years
  TTP
Part 1 - To assess preliminary antitumor activity of LOXO-338 based on duration of response (DOR) | Estimated up to 2 years
  DOR
Part 2 - To characterize the pharmacokinetics (PK) properties of LOXO-338 in combination with pirtobrutinib: Area under the plasma concentration versus time curve (AUC) | Predose up to 24 hours postdose
  PK: AUC of LOXO-338 alone and in combination with pirtobrutinib
Part 2 - To characterize the PK properties of LOXO-338 and in combination with pirtobrutinib: Maximum drug concentration (Cmax) | Predose up to 24 hours postdose
  PK: Cmax of LOXO-338 alone and in combination with pirtobrutinib
Part 2 - To assess preliminary antitumor activity of LOXO-338 alone and in combination with pirtobrutinib based on overall response rate (ORR) | Estimated up to 2 years
  ORR
Part 2 - To assess preliminary antitumor activity of LOXO-338 alone and in combination with pirtobrutinib based on progression-free survival (PFS) | Estimated up to 2 years
  PFS
Part 2 - To assess preliminary antitumor activity of LOXO-338 alone and in combination with pirtobrutinib based on time-to-progression (TTP) | Estimated up to 2 years
  TTP
Part 2 - To assess preliminary antitumor activity of LOXO-338 alone and in combination with pirtobrutinib based on duration of response (DOR) | Estimated up to 2 years
  DOR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- United States (13):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California San Francisco, Medical Center at Paranassus, San Francisco, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana Blood & Marrow Transplantation (IBMT), Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (6):
  - L'Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse, Cedex 9
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Cedex
  - CHRU de Montpellier-Hopital St Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Institut Curie, Paris
  - Centre hospitalier universitaire de Haut Leveque, Pessac
- IRCCS - AOU di Bologna, Bologna, Italy
- Poland (3):
  - Centrum Medyczne Pratia Poznan, Skorzewo, Poznan
  - Pratia MCM Krakow, Krakow
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwiatek M, Murthy GSG, Hoffmann M, Tessoulin B, Danilov A, Alencar AJ, Shah NN, Ghesquieres H, Le Gouill S, Jurczak W, Han H, Yuen E, Patel V, Guo-Avrutin Y, Pauff JM, Roeker LE. A First-in-Human Phase I Study of LOXO-338, an Oral Selective Bcl-2 Inhibitor, in Patients With Advanced Hematologic Malignancies. Clin Lymphoma Myeloma Leuk. 2025 Jul;25(7):512-519. doi: 10.1016/j.clml.2025.01.018. Epub 2025 Jan 28. PMID 40000354
- See also: Study of Oral LOXO-338 in Patients with Advanced Blood Cancers — https://trials.lillytrialguide.com/en-US/trial/3WoOdectArUAmQZPkKcclh?nickname=J3N-OX-JZRA